CLINICAL TRIAL: NCT06934538
Title: Open Label, Multicenter, Dose-escalation and Cohort-expansion Phase I/IIA Trial of STC-1010, an Immunotherapy, in Patients With Unresectable Locally Advanced or Metastatic Colorectal Cancer (CRC) - BreAK CRC Trial (BreAK for Brenus Anti-cancer)
Brief Title: First-in-human Trial of STC-1010, an Immunotherapy, in Patients With Unresectable Locally Advanced or Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brenus Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BreAK CRC-001
Record Dates: First submitted 2024-05-16; First posted 2025-04-18 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-07

CONDITIONS: Unresectable Metastatic Colorectal Cancer; Unresectable Locally Advanced Colorectal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Phase 1 (Experimental): Dose-escalation and small expansion study in BRAF wild type, KRAS mutated, unresectable stage IIIC (T4b) or unresectable stage IV CRC participants with microsatellite stable (MSS) disease who have not received prior treatment
  Interventions: Biological: STC-1010 + IS regimen + SOC therapy
- Phase 2A: Arm 2A-1 (Experimental): Evaluation of safety and efficacy in BRAF wild type, KRAS mutated, unresectable stage IIIC (T4b) or unresectable stage IV CRC participants with MSS disease
  Interventions: Biological: STC-1010 + IS regimen + SOC therapy
- Phase 2A: Arm 2A-2 (Experimental): Evaluation of safety and efficacy in BRAF wild type, KRAS mutated, unresectable stage IIIC (T4b) or unresectable stage IV CRC participants with microsatellite instability-high (MSI-H) disease
  Interventions: Biological: STC-1010 + IS regimen + SOC therapy

INTERVENTIONS:
Biological: STC-1010 + IS regimen + SOC therapy — STC-1010 administered with immunostimulants (IS) in low-dose (cyclophosphamide and GM-CSF) and standard of care (SOC) therapy (mFOLFOX6 with or without bevacizumab)

SUMMARY:
This is a phase I/IIA, first-in-human (FIH), two-part, open-label, multicenter study to characterize the safety, tolerability profile, and clinical efficacy of STC-1010 associated with GM-CSF and cyclophosphamide immunostimulant (IS) regimen administered with standard of care (SOC) therapy (mFOLFOX6 with or without bevacizumab) to participants with unresectable locally advanced (stage IIIC, T4b) or unresectable metastatic (stage IV) colorectal cancer (CRC).

The trial will be conducted in two parts:

* A Phase I consisting of a dose escalation part and small expansion part to determine the maximum tolerated dose (MTD), recommended Phase II dose (RP2D) and safety profile of the STC-1010 + IS regimen administered with SOC therapy. Approximately 21 to 33 participants will be included in this phase in Europe.
* A Phase IIA consisting of the expansion stage of the study which will further evaluate the clinical efficacy and safety of STC-1010 on a larger number of participants treated at the identified RP2D. Approximately 57 to 60 participants will be enrolled in total in 2 different arms. Multi-site recruitment will take place in Europe and in the US.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-75 years
2. Histologically confirmed diagnosis of unresectable locally advanced (stage IIIC, T4b) or unresectable metastatic (stage IV) (R0) adenocarcinoma of the colon or rectum
3. Adjuvant fluoropyrimidine monotherapy or oxaliplatin-based chemotherapy allowed if more than 6 months have elapsed between the end of adjuvant treatment and first relapse
4. Determination of KRAS and BRAF mutation status
5. Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
6. Must agree to have biopsy at screening and on-treatment, only if not representing an unacceptable clinical risk and/or if technically feasible as judged by the Investigator in discussion with the interventional radiologist or endoscopist
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1. Participants >70 years must have a PS= 0.
8. Life expectancy > 3 months as assessed by the investigator
9. Effective contraceptive measures implemented

Exclusion Criteria:

1. Patients with symptomatic ascites or pleural effusion
2. Dihydropyrimidine dehydrogenase (DPD) deficiency
3. Resectable tumor with curative intent or patient considered for a curative strategy by intensifying chemotherapy to induce resectability
4. Prior chemotherapy for metastatic disease
5. Prior immunotherapy for advanced/metastatic disease (except for Arm 2A-2)
6. Prior therapy with an investigational agent
7. BRAF mutation
8. Active auto-immune diseases such as rheumatoid arthritis, lupus, Crohn's disease, ulcerative colitis
9. Medical conditions requiring immunosuppressive therapy
10. Major surgery <4 weeks prior to first administration of STC-1010
11. Radiotherapy < 4 weeks prior to first administration of STC-1010 or < 2 weeks in case of palliative radiotherapy
12. Prior stem cell or solid organ transplantation
13. Dementia or altered mental status or subject of a legal protection measure that would prohibit informed consent
14. Active drug or alcohol abuse as assessed by the Investigator
15. Participant deprived of their liberty by a judicial or administrative decision, undergoing psychiatric care and admitted to a health or social establishment for purposes other than research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1: To determine overall safety profile, recommended Phase 2 dose (RP2D) and maximum tolerated dose (MTD) | 28 days
  Endpoint/Outcome Measures:
  Incidence, severity, and relationship of Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Dose-Limiting Toxicities (DLT) (in dose escalation part), AEs leading to treatment discontinuation; and clinically significant findings on clinical laboratory tests, vital signs, electrocardiograms (ECGs), and physical examinations, using the Common Terminology Criteria for Adverse Events (CTCAE Version 5).
Phase 2A: To determine the clinical efficacy by Progression Free Survival (PFS) rate | 12 months
  Progression Free Survival (PFS) rate at 12 months from STC-1010 + IS regimen initiation, defined as the proportion of participants alive and without progression (i.e., participants with complete response [CR], partial response [PR] or stable disease [SD]) at 12 months according to RECIST 1.1

SECONDARY OUTCOMES:
Phase 1: To determine the preliminary clinical efficacy | 6 months
  Endpoints/Outcome Measures: Overall Response Rate (ORR) at 6 months from STC-1010 + IS treatment initiation, defined as the achievement of either a complete response (CR) or partial response (PR) according to RECIST 1.1; Progression Free Survival (PFS) rate at 6 months from STC-1010 + IS treatment initiation (defined as the rate of participants alive with CR, PR or SD) according to RECIST 1.1; and Median of PFS.
Phase 1: To describe the effects on cell-mediated immunity | Up to 72 hours post injection
  Assessment of delayed-type hypersensitivity (DTH) score after the first vaccination (at 1, 24, 48 and 72 hours post-STC-1010 injection) and then after the 4th, 8th and every boost
Phase 2A: To determine the overall safety and tolerability profile | 6, 12 and 24 months
  Endpoints/Outcome Measures: Incidence, severity and relationship of TEAEs, SAEs, TEAEs leading to discontinuation of study treatment; and clinically significant findings on clinical laboratory tests, vital signs, ECGs and physical examinations, using the CTCAE Version 5.
Phase 2A: To determine the clinical efficacy by Clinical Benefit Rate (CBR) | 12 and 24 months
  Clinical Benefit Rate (CBR) defined as the percentage of participants in whom the best response is CR or PR, or SD lasting for a least 6 months.
Phase 2A: To determine the clinical efficacy by Objective Response Rate (ORR) | 6, 12 and 24 months
  Objective Response Rate (ORR) defined as the proportion of patients who achieve a complete or partial response per RECIST 1.1 criteria. Patients with unevaluable or unknown response status will be considered as non-responders.
Phase 2A: To determine the clinical efficacy by Duration of Response (DOR) | 6,12 and 24 months
  Duration of response (DOR), defined as the time from first documented evidence of CR or PR to the earliest date of documented radiological progression or death due to any cause
Phase 2A: To determine the clinical efficacy by Progression Free Survival (PFS) | 6,12 and 24 months
  Progression Free Survival (PFS) defined as the time to the date of progression or death from any cause. The median PFS with it's 95% confidence interval (CI) will also be calculated
Phase 2A: To determine the clinical efficacy by Overall Survival (OS) | 12 and 24 months
  Overall Survival (OS) defined as the time to the date of death from any cause. The median OS with its 95% CI will also be calculated.
Phase 2A: To determine the clinical efficacy by metastases resection rate | Up to 18 months
  Metastases resection rate defined as the percentage of participants who undergo resection

OTHER OUTCOMES:
Phase 1: To determine the impact on immune and molecular biomarkers (exploratory outcomes) | At baseline/screening (T0), 1 month, 2 months, 6 months, 12 months
  Assessment of biomarkers in blood and tumor biopsies
Phase 2: To determine the impact on immune and molecular biomarkers (exploratory outcomes) | At baseline/screening (T0), 1 month, 2 months, 6 months, 12 months and at time of progression (Tprogression, up to 24 months)
  Assessment of biomarkers in blood and tumor biopsies

CONTACTS AND LOCATIONS:
Locations (9):
- Johns Hopkins, Baltimore, Maryland, United States
- Institut Jules Bordet, Brussels, Belgium
- France (7):
  - Institut Bergonié, Bordeaux
  - Centre Georges François Leclerc (CGFL), Dijon
  - Centre Léon Bérard (CLB), Lyon
  - Hospices Civils de Lyon (HCL), Lyon
  - Institut du Cancer de Montpellier (ICM), Montpellier
  - Centre Hospitalier Universitaire de Poitiers (CHU), Poitiers
  - Institut Gustave Roussy (IGR), Villejuif

IPD SHARING:
Plan to Share IPD: Undecided